CLINICAL TRIAL: NCT00069927
Title: Adderall-XR Versus Concerta For Cancer Treatment-Related Neurocognitive Sequelae And Depression In Pediatric Patients: A Randomized Phase II Study
Brief Title: Adderall XR Compared With Concerta in Treating Young Cancer Patients With Memory, Attention, and Depression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Only 12 subjects enrolled. DSMB recommended closing due to lack of feasibility
Sponsor: University of South Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: SCUSF 0201; HLMCC-0201 (Other: H. Lee Moffitt Cancer Center Research Base); U10CA081920 (NIH); SCUSF-0201 (Other: SunCoast CCOP Research Base)
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Depression; Neurotoxicity; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific; depression; neurotoxicity
MeSH Terms: conditions — Depression; Neurotoxicity Syndromes | interventions — SLI381; Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1- Adderall- XR® (Experimental): Adderall-XR® 1 10 mg/day for 3-12 weeks depending on subject's response
  Interventions: Drug: Adderall-XR®; Drug: Concerta®
- Arm II Concerta® (Experimental): Concerta ® 18 mg/day for 3-12 weeks depending on subject's response
  Interventions: Drug: Adderall-XR®; Drug: Concerta®

INTERVENTIONS:
Drug: Adderall-XR® — Adderall-XR® 10 mg/day for 3-12 weeks depending on subject's response
  Other Names: dextroamphetamine-amphetamine
Drug: Concerta® — Concerta® 18 mg/day for 3-12 weeks depending on subject's response
  Other Names: methylphenidate hydrochloride

SUMMARY:
RATIONALE: Stimulant drugs such as dextroamphetamine-amphetamine and methylphenidate may help improve memory, attention, and thinking problems caused by central nervous system (CNS) treatment for cancer, and may help decrease depression.

PURPOSE: This randomized phase II trial is studying dextroamphetamine-amphetamine to see how well it works compared to methylphenidate in treating depression and problems with memory, attention, and thinking in children who have undergone CNS treatment for cancer. This trial will also study how often depression is seen and if these medications might help.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the response rates in pediatric cancer patients with treatment-related neurocognitive sequelae treated with dextroamphetamine-amphetamine (Adderall-XR®) vs methylphenidate (Concerta®).
* Compare the durability of response at 12 weeks in patients who show a response at 3 weeks after treatment with these drugs.
* Determine whether patients who have no response to one of these study drugs can respond to the other study drug.
* Determine the prevalence of depression and possible response to neurostimulant therapy in this patient population.

OUTLINE: This is a randomized, multicenter study.

Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral dextroamphetamine-amphetamine once daily for 3 weeks. Patients who achieve response (based on neurocognitive testing) continue treatment for a total of 12 weeks. Patients with no response after 3 weeks cross over to arm II after a 48-hour washout period.
* Arm II: Patients receive oral methylphenidate once daily for 3 weeks. Responding patients continue treatment for a total of 12 weeks. Patients with no response after 3 weeks cross over to arm I after a 48-hour washout period.

Depression and neurocognitive function are assessed at baseline, 3 weeks, and end of study.

PROJECTED ACCRUAL: A total of 177 patients (approximately 88 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
INCLUSION CRITERIA:

* Between the ages of 6-17 at the time of study participation.
* Have a diagnosis of any malignancy that required CNS treatment such as surgery and/or irradiation and/or intrathecal chemotherapy. (Patients treated with systemic chemotherapy alone are not eligible to participate)
* Off treatment and cancer free for a minimum of 6 months.
* Have a proficiency in English.

EXCLUSION CRITERIA:

* Patients with an estimated intelligence quotient (IQ) of less than 65 (based on the Wide Range Achievement Test (WRAT-3) Reading subtest) are not eligible to continue on study.
* At least one standard deviation below the level of performance predicted by their IQ on at least 2 of the 3 WISC-III subtests.
* Diagnosed with Attention Deficit Disorder (ADD) or Attention Deficit Hyperactivity Disorder (ADHD) prior to their cancer diagnosis.
* Currently taking antidepressants, antipsychotics, or other stimulants.
* Are blind.
* Have glaucoma.
* Family history of motor and phonic tics or Tourette's syndrome.
* Have seizures not controlled by antiepileptic drugs. (Note: Patients who are not experiencing seizure activity, having been on a stable dose of an antiepileptic drug for at least 12 weeks may participate)
* Taking a monoamine oxidase (MAO) inhibitor.
* Have a history of cardiovascular disease, uncontrolled hypertension or hyperthyroidism.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2003-08; Primary Completion 2006-06 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Response rate as measured by Wechsler Intelligence Scale for Children-III (WISC III) subtest: Coding, Symbol Search and Digit Span at baseline, and 3 weeks after the start of study treatment | 12 weeks

SECONDARY OUTCOMES:
Durability of response as measured by WISC III subtest: Coding, Symbol Search and Digit Span at 12 weeks after the start of study treatment | 12 weeks
Depression as measured by Children's Depression Inventory Short Version (CDI-S) at baseline, weeks 3 and 12 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Booth-Jones, PhD, Study Chair — University of South Florida
Locations (9):
- United States (9):
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Sacred Heart Children's Hospital, Pensacola, Florida
  - St. Joseph's Children's Hospital of Tampa, Tampa, Florida
  - CCOP - Florida Pediatric, Tampa, Florida
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - CHRISTUS Santa Rosa Children's Hospital, San Antonio, Texas
  - MBCCOP - South Texas Pediatrics, San Antonio, Texas